CLINICAL TRIAL: NCT04201990
Title: An Exploratory Study on the Safety and Efficacy of Cryoablation Combined With Camrelizumab and Apatinib in the Treatment of Multiprimary Lung Cancer With Non-known Driving Genes
Brief Title: Cryoablation Combined With Camrelizumab and Apatinib for Multiprimary Lung Cancer
Acronym: CCA-MPLC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ShiYue Li (Other)
Responsible Party: Sponsor-Investigator, ShiYue Li, Deputy Director of Guangzhou Institute of Respiratory Disease, Guangzhou Institute of Respiratory Disease
Organization: Guangzhou Institute of Respiratory Disease (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-62
Record Dates: First submitted 2019-12-03; First posted 2019-12-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Lung Cancer
Keywords: MPLC; Camrelizumab; Apatinib
MeSH Terms: conditions — Lung Neoplasms | interventions — camrelizumab; apatinib; Cryosurgery

STUDY DESIGN:
Intervention Model Description: About two to three weeks after cryoablation, Eligible patients sign informed consent and then begin treating with Camrelizumab and Apatinib.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): Camrelizumab, iv, Q3W until progression disease or intolerable toxicity or 2 years Apatinib, po, QD until progression disease or intolerable toxicity or 2 years
  Interventions: Drug: Camrelizumab and Apatinib

INTERVENTIONS:
Drug: Camrelizumab and Apatinib — Camrelizumab, iv, Q3W; Apatinib, po, QD
  Other Names: cryoablation

SUMMARY:
Objective: This study is to observe the safety and therapeutic effect of cryoablation combined with pd-1 antibody immunotherapy and anti-angiogenesis therapy in multiple primary lung cancer (MPLC) patients.

Methods: In this study, 20 patients with MPLC who conform to the admission criteria are enrolled and began to receive treatment with Camrelizumab combined with Apatinib after cryoablation.

DETAILED DESCRIPTION:
Subjects who meet the admission criteria will be treated with Camrelizumab and Apatinib until disease progression, intolerable toxicity, death, withdrawal of the patient or the researchers determined that the drug must be discontinued.

The primary end point of this study is safety of cryoablation combined with carillizumab and apatinib for MPLC. The secondary endpoints include objective response rate, disease control rate, time to progression, progression free survival and overall survival. Exploratory endpoint is to explore biomarkers in tumor tissue and blood that could potentially predict the efficacy of Camrelizumab and Apatinib.

ELIGIBILITY:
Inclusion Criteria:

1. clinical and pathological diagnosis of muitiple primary lung cancer.
2. more than three pulmonary nodules and without lymph node metastasis.
3. the maximum lesion less than three centimeters in diameter.
4. No more than one operation, and remains more than two pulmonary nodules which pathological confirmed were MIA or AIS.
5. at least one measurable lesion conforming to RECIST v1.1 standard was left after cryotherapy.
6. male or female, age 18 to 75 years old.
7. the ECOG PS score was 0 or 1.
8. expected survival is more than 12 weeks.
9. functions of vital organs and bone marrow meet the following requirements: A. ANC ≥1.5× 109/L, PLT ≥100× 109/L, HGB ≥9 g/dL; B. TBIL ≤1.5 ULN, ALT and/or AST ≤2.5 ULN, ALB ≥2.8 g/dL; C. Cr ≤1.5× ULN, or creatinine clearance rate ≥40 mL/min
10. subject and subject's sexual partner shall use a medically approved contraceptive method during the study treatment period and within 6 months after the end of the study treatment period.
11. subject must sign theinformed consent.

Exclusion Criteria:

1. patients with EGFR mutations and ALK rearrangement.
2. cannot be treated with cryoablation: diffuse lesions in both lungs, extensive pleural metastasis with large amount of pleural effusion, tumor adjacent to mediastinal large vessels or surrounding large vessels.
3. have previously received anti-pd-1, anti-pd-l1, anti-ctla-4 antibodies or any other antibodies or drugs that target T cell co-stimulation or immune checkpoint pathways.
4. received the following treatment Within four weeks before enrollment:

   * received systemic anti-tumor therapy, such as chemotherapy, targeted therapy and immunotherapy;
   * receive any investigational medication;
   * receive a large dose of immunosuppressive drugs (systemic glucocorticoid exceeding 10 mg/ temprednisone or its equivalent);
   * receive live attenuated vaccine;
   * major surgery or unhealed surgical wounds, ulcers, or fractures.
5. known or suspected active autoimmune diseases (congenital or acquired).
6. allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation.
7. allergy to any component of monoclonal antibody preparation.
8. interstitial lung disease.
9. suffering from other uncontrolled serious diseases, including but not limited to:

   * severe infections in the active phase or with poor clinical control;
   * HIV infection (HIV antibody positive);
   * acute or chronic active hepatitis B (HBV DNA positive) or acute or chronic active hepatitis C (HCV antibody positive);
   * active tuberculosis;
   * grade iii-iv congestive heart failure (New York cardiology association classification), poorly controlled and clinically significant arrhythmia;
   * uncontrolled arterial hypertension (systolic blood pressure ≥160mmHg or diastolic blood pressure ≥100mmHg);
   * any arterial thrombosis, embolism or ischemia, such as myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack, occurred within 6 months;
   * diseases requiring anticoagulant therapy with farfarin (coumarin);
   * uncontrolled hypercalcemia or symptomatic hypercalcemia requiring continued bisphosphate therapy;
   * accompanied by other malignant tumors (except those that have been cured, such as carcinoma in situ of the cervix, non-melanoma skin cancer, etc.).

     10. The participants were judged to be unsuitable for the study by investigator.

     11. Pregnant or nursing women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Safety score | three weeks
  The occurrence of grade 3 to 5 adverse reactions was assessed by CTC AE v5.0

SECONDARY OUTCOMES:
ORR | six weeks
  objective response rate
DCR | six weeks
  Disease control rate
PFS | six weeks
  progression free survival
OS | six weeks
  Overall survival
DOR | six weeks
  Duration of response

OTHER OUTCOMES:
biomarker | three months
  To explore biomarkers in tumor tissue and blood that could potentially predict the efficacy of Camrelizumab and Apatinib like PD-L1, ctDNA, CEA， CA125， CA153.